CLINICAL TRIAL: NCT05393596
Title: Effects of Virtual Reality Software on Levels of Stigma Towards People With Mental Illness: An Experimental Study.
Brief Title: Effects of Virtual Reality Software on Levels of Stigma Towards People With Mental Illness.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Desarrollo (Other)
Responsible Party: Principal Investigator, Matías E. Rodríguez-Rivas, Principal Investigator, Universidad del Desarrollo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 513
Record Dates: First submitted 2022-05-18; First posted 2022-05-26 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Social Stigma; Virtual Reality
Keywords: Stigma; Virtual Reality; Randomized Control Trial
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Incluyete VR Software) (Experimental): Through virtual reality headsets, the software Inclúyete VR will be used, in which situations related to stigma in Severe Mental Disorder are recreated. Specifically, its purpose is to put the participant in a virtual world that shows how the stigma towards people with severe mental health problems is and also to experience situations of rehabilitation and social inclusion, thus giving a more real and closer image of what can be the current treatment in mental health. The approximate duration is 15 minutes.
  Interventions: Behavioral: Virtual Reality Software Intervention
- Control Group (Welcome Oculus Software) (Active Comparator): Participants will use the default virtual reality headset welcome game, unrelated to mental health. It presents an interactive virtual environment, with various playful interfaces and instructions for use. The duration is approximately 15 minutes.
  Interventions: Behavioral: Virtual Reality Software Intervention

INTERVENTIONS:
Behavioral: Virtual Reality Software Intervention — Virtual Reality Software Intervention

SUMMARY:
The purpose of the research is to contribute to the reduction of stigma among university students among people with serious psychiatric illnesses and to improve future educational processes focused on the social inclusion of people with these mental health problems.

For this purpose, the methodology proposed is a mixed (qualitative and quantitative), with an experimental design. Students of the Universidad del Desarrollo will be contacted and invited to participate voluntarily, after signing an informed consent of the research. This procedure will consist of the use of a virtual reality software in the university premises, together with the application of a survey with scales validated in Chile before and after the intervention, in addition to a semi-structured interview about the experience in the use of the software, together with the identification of strengths and opportunities for improvement of the intervention. The total estimated duration of the procedure is approximately 35 minutes.

It is expected to determine the level of stigma towards mental illness before and after the development of the virtual reality intervention, in addition to describing the perception of the students' experience after participating in the intervention (including an analysis of strengths and opportunities for improvement).

The general objective of the present research is to evaluate the effect of a virtual reality intervention on levels of stigma towards people with mental illness in university students.

DETAILED DESCRIPTION:
Stigma towards people with mental illness represents a serious public health problem worldwide and is considered the main barrier in the social inclusion and participation of affected people, which has a negative impact on their quality of life, determining even a higher risk of suicide and mortality, along with a lower life expectancy compared to the unaffected population.

Faced with the high levels of stigmatization present in society, several initiatives and studies have been conducted worldwide focused on its reduction, where it has been shown that direct contact with people with psychiatric illnesses and education are key and effective interventions, especially when conducted and focused on strategic groups, such as professionals and students in training.

Despite the fact that direct contact and activities in which participants and users share thoughts and experiences around mental health have been shown to be key to the success of these programs, their implementation in virtual learning spaces is recent, particularly for university students.

Thus, several authors have shown that innovative interventions using new technologies, such as the use of video games, the application of virtual reality, the use of simulated actors and e-contact through virtual media with mental health users, are effective tools in developing various skills, tools and fostering an inclusive attitude with a focus on reducing prejudice and stigma towards individuals with severe mental disorders.

Despite this, there is currently a gap in knowledge about the effects of virtual reality programs focused on decreasing stigma towards people with psychiatric illnesses.

General objective: To evaluate the effect of a virtual reality intervention on levels of stigma toward people with mental illness in university students.

Specific objectives:

1. To measure the level of stigma toward people with mental illness of students pre- and post-participation in the virtual reality intervention
2. To describe students' perception of the experience after participating in the virtual reality intervention.
3. To identify strengths and opportunities for improvement in the virtual reality intervention.

In order to achieve the proposed objectives, a mixed methodology (qualitative and quantitative) will be used in a randomized experimental design. The population will be composed of undergraduate students of the Universidad del Desarrollo, and the sampling technique will be non-probabilistic by convenience.

The inclusion criteria are described as: a) age over 18 years; b) being an undergraduate or postgraduate student at Universidad del Desarrollo; c) having signed the full or abbreviated informed consent form.

The sample will be composed of 100 students, who will be randomized into the following control and experimental groups:

1. Control group: Participants will use the default virtual reality headset welcome game, unrelated to mental health. It presents an interactive virtual environment, with various playful interfaces and instructions for use. The duration is approximately 15 minutes.
2. Experimental group: The software Inclúyete VR will be used, in which situations related to stigma in Severe Mental Disorder are recreated. Specifically, its purpose is to put the participant in a virtual world that shows how the stigma towards people with severe mental health problems is and also to experience situations of rehabilitation and social inclusion, thus giving a more real and closer image of what can be the current treatment in mental health. The approximate duration is 15 minutes.

Stigma levels will be evaluated before and after the intervention in the experimental and control groups, through the application of the following scales validated in Spanish in Chile: a) Attribution Questionnaire AQ-27, b) Questionnaire on Student Attitudes toward Schizophrenia. The application of these instruments will be done in a Google form through a tablet of the research team, which includes the abbreviated informed consent. The total estimated time to respond is approximately 10 minutes.

Along with this, a semi-structured recorded interview will be conducted with the participants of the experimental group, with an estimated duration of 10 minutes. The collection of qualitative data about the experience in changing the stigma towards mental illness, together with the identification of strengths and opportunities for improvement of the intervention will be carried out through a recorded semi-structured interview, using the following script of questions:

1. How do you evaluate the experience of the virtual reality intervention in terms of its usefulness and/or potential benefits in the social inclusion of people with psychiatric illnesses?
2. What were the main learnings and knowledge acquired during the intervention?
3. How could I incorporate those learnings and knowledge into my role as a student and future professional in terms of social inclusion of people with mental health problems?
4. Did your perception of inclusion of people with psychiatric illnesses change? In what way?
5. What are the main strengths and positive aspects of the software?
6. What do you think are the main weaknesses or aspects to be improved in future instances and versions of the software?

Finally, participants will have the option of allowing themselves to be contacted via e-mail to answer a follow-up survey through a Google questionnaire, which will be carried out 4 weeks after the application of the study.

Data analysis will be performed using NVivo V.11 software for content analysis of the qualitative data, and SPSS software for descriptive statistics in relation to the quantitative data.

Ethical considerations:

From the point of view of the principle of autonomy, student participation in this research project is free and voluntary. Regarding the principles of beneficence and non-maleficence, the way the research is designed, it does not entail any risk or expense for the students. Neither will the students benefit directly from the results obtained; however, answering the scales and participating in the semi-structured interview will contribute to improve future educational and research instances. Refusal to participate, or withdrawal from the study at any time, does not alter any aspect of the student's relationship with the University, and has no present or future influence on the student's academic performance. In relation to the principle of fairness, all undergraduate students at Universidad del Desarrollo will have the same opportunity to participate in the study.

Ethical Considerations for Personal Data Protection and Confidentiality:

The answers to the scales obtained through Google forms will be anonymous. All of them will be analyzed after assigning them a numerical code, so there is no risk of disclosing identifying information of any student, such as name, e-mail, etc. All scales will be downloaded to the institutional computer of the responsible researcher, and will be stored for the duration of the research. Once the research is concluded, all stored information will be destroyed and discarded. Regarding the semi-structured interview, it will be recorded and identified with an assigned numerical ID, which allows anonymizing the students, with the aim of facilitating the subsequent transcription and content analysis of the stories.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Being an undergraduate or postgraduate student at Universidad del Desarrollo

Exclusion Criteria:

- Participants who have not signed the full or abbreviated informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in stigma levels pre- and post-intervention. | Pre intervention and immediately post intervention
  Stigma levels will be evaluated in the experimental and control groups, pre- intervention and immediately after the intervention of the Virtual Reality Software, through the measurement of the following scale validated in Spanish:
  a) Attribution Questionnaire AQ-27
Changes in stigma levels pre- and post-intervention. | Pre intervention and immediately post intervention.
  Stigma levels will be evaluated in the experimental and control groups, pre- intervention and immediately after the intervention of the Virtual Reality Software, through the measurement of the following scale validated in Spanish:
  b) Questionnaire on Student Attitudes toward Schizophrenia.

SECONDARY OUTCOMES:
Qualitative perception of the experience, strengths and opportunities to improve the software, after participating in the Virtual Reality Experimental group intervention (Inclúyete VR). | Immediately post intervention
  A semi-structured recorded interview will be conducted with the participants of the experimental group (Inclúyete VR). The collection of qualitative data will be carried using the following script of questions:
  1. How do you evaluate the experience of the virtual reality intervention in terms of its usefulness and/or potential benefits in the social inclusion of people with psychiatric illnesses?
  2. What were the main learnings and knowledge acquired during the intervention?
  3. How could I incorporate those learnings and knowledge into my role as a student and future professional in terms of social inclusion of people with mental health problems?
  4. Did your perception of inclusion of people with psychiatric illnesses change? In what way?
  5. What are the main strengths and positive aspects of the software?
  6. What do you think are the main weaknesses or aspects to be improved in future instances and versions of the software?

CONTACTS AND LOCATIONS:
Overall Officials: Matías E. Rodríguez-Rivas, Principal Investigator — Universidad del Desarrollo
Locations (1):
- Universidad del Desarrollo, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez-Rivas ME, Cangas AJ, Fuentes-Olavarria D. Controlled Study of the Impact of a Virtual Program to Reduce Stigma Among University Students Toward People With Mental Disorders. Front Psychiatry. 2021 Feb 9;12:632252. doi: 10.3389/fpsyt.2021.632252. eCollection 2021. PMID 33633613
- [Background] Yuen ASY, Mak WWS. The Effects of Immersive Virtual Reality in Reducing Public Stigma of Mental Illness in the University Population of Hong Kong: Randomized Controlled Trial. J Med Internet Res. 2021 Jul 14;23(7):e23683. doi: 10.2196/23683. PMID 34259636
- [Background] Cangas AJ, Galván B. Estudio preliminar de la utilidad de un programa de realidad virtual contra el estigma en salud mental. Rev INFAD Psicol Int J Dev Educ Psychol. 2020;1(1):45-52. doi:10.17060/ijodaep.2020.n1.v1.1760
- [Background] Rodriguez-Rivas ME, Cangas AJ, Cariola LA, Varela JJ, Valdebenito S. Innovative Technology-Based Interventions to Reduce Stigma Toward People With Mental Illness: Systematic Review and Meta-analysis. JMIR Serious Games. 2022 May 30;10(2):e35099. doi: 10.2196/35099. PMID 35635744
- [Derived] Rodriguez-Rivas ME, Cangas AJ, Martin A, Romo J, Perez JC, Valdebenito S, Cariola L, Onetto J, Hernandez B, Ceric F, Cea P, Corrigan P. Reducing Stigma Toward People with Serious Mental Illness Through a Virtual Reality Intervention: A Randomized Controlled Trial. Games Health J. 2024 Feb;13(1):57-64. doi: 10.1089/g4h.2023.0118. Epub 2023 Sep 11. PMID 37695822